CLINICAL TRIAL: NCT01132742
Title: Malnutrition and Outcome in Hospitalized Children in Europe (ESPEN Network Grant Project)
Brief Title: Malnutrition and Outcome in Hospitalized Children in Europe
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Koletzko - Office, Prof, Ludwig-Maximilians - University of Munich
Other Study IDs: ESPEN
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Malnutrition
Keywords: Malnutrition; children; Hospital Stay; Screening Tools; Anthropometry
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- hospitalised children

SUMMARY:
Malnutrition in children has even more severe consequences on disease course and long-term health than malnutrition in adults. According to prior studies, malnutrition affects about 15-30 % of hospitalized children in Europe (ESPGHAN 2005, Pawellek et al 2008, Joosten and Hulst 2008). However, available criteria for defining malnutrition in paediatric patients are inconsistent, not based on firm evidence, and not generally agreed upon. Current guidelines do not address assessment of and screening for childhood malnutrition. Therefore, a large number of affected children are not adequately diagnosed.

One aim of this study is to assess the prevalence of malnutrition and patients at risk for malnutrition among at least 2700 hospitalized children mainly across Europe. In addition criteria to link anthropometric measurements and the prediction of outcome, i.e. length of hospital stay, shall be established. A further goal then is to establish agreed, evidence-based criteria for malnutrition in children with the purpose of leading to an agreed, evidence-based screening tool for paediatric malnutrition in developed countries. This tool shall include a set of simple questions, based on previously suggested tools. Thereby this study will provide a strong basis for implementing evidence-based nutritional interventions in paediatric patients by harmonisation of diagnostic criteria for childhood malnutrition in developed countries.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted to the participating hospitals during the study period
* Age between 1 month and 18 years
* Expected hospital stay exceeding 24 hours
* Parents/caregivers, as well as those patients capable to comprehend, agree to participation and sign the informed consent form

Exclusion Criteria:

* Infants with premature birth (<37 weeks gestational age) during the first 12 months of life
* Infants < 1 month of age
* Patients ≥ 18 years of age
* Children in need of intensive care
* Children admitted to day-care (LOS < 24hours)
* Patients admitted for elective reasons with an expected hospital stay <24 hours

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will be performed in hospitalized children attending general paediatric wards. The network comprises at least 13 teams from at least 11 countries. A total of 2700 patients will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 2567 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | 60 days
  Length of Hospital Stay will be compared between malnourished and non malnourished children.

SECONDARY OUTCOMES:
infection as a complication during hospital stay | 60 days
  frequency of infectious complications (number of days with temperature >38,5°C, number of days with days with antibiotic use)
gastrointestinal complications (vomiting, diarrhoea) | 60 days
  frequency of gastrointestinal complications: frequency of vomiting and diarrhoea during hospital stay
muscle strength | within 24 hours after admission
  maximal isometric grip force in children ≥ 6 years of age measured within 24 hours after admission

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (14):
- Children's Hospital Zagreb, Zagreb, Croatia
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark
- Paediatric Clinical Investigation Center Unit (CIC-9301-Inserm-CHU) and U995-Inserm, hospital Jeanne de Flandre, University hospital of Lille., Lille, France
- Dr. von Hauner Children's Hospital. Munich, Germany, Munich, Bavaria, Germany
- Technological Education Institute, Thessaloniki, Greece
- Schneider Children's Hospital, Petah Tikvah, Israel
- Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico - Milano, Milan, Italy
- Netherlands (2):
  - Beatrix Children's Hospital, University Medical Center Groningen, Groningen
  - Sophia Children's Hospital, Erasmus University, Rotterdam
- Poland (2):
  - Medical Univ. of Warsaw, Warsaw
  - The Children's Memorial Health Institute, Warsaw
- Spitalul Clinic da Urgenta pentru Copii, Cluj-Napoca, Romania
- United Kingdom (2):
  - Oxford Children's Hospital, Oxford
  - Royal Hospital for Sick Children, Yorkhill Glasgow

REFERENCES:
- [Derived] Chourdakis M, Hecht C, Gerasimidis K, Joosten KF, Karagiozoglou-Lampoudi T, Koetse HA, Ksiazyk J, Lazea C, Shamir R, Szajewska H, Koletzko B, Hulst JM. Malnutrition risk in hospitalized children: use of 3 screening tools in a large European population. Am J Clin Nutr. 2016 May;103(5):1301-10. doi: 10.3945/ajcn.115.110700. Epub 2016 Apr 20. PMID 27099244
- [Derived] Hecht C, Weber M, Grote V, Daskalou E, Dell'Era L, Flynn D, Gerasimidis K, Gottrand F, Hartman C, Hulst J, Joosten K, Karagiozoglou-Lampoudi T, Koetse HA, Kolacek S, Ksiazyk J, Niseteo T, Olszewska K, Pavesi P, Piwowarczyk A, Rousseaux J, Shamir R, Sullivan PB, Szajewska H, Vernon-Roberts A, Koletzko B. Disease associated malnutrition correlates with length of hospital stay in children. Clin Nutr. 2015 Feb;34(1):53-9. doi: 10.1016/j.clnu.2014.01.003. Epub 2014 Jan 11. PMID 24461472